#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a randomized open-label relative bioavailability study to compare the pharmacokinetic parameters of a lower dose formulation of ambrisentan (GSK1325760) with marketed ambrisentan in healthy adult participants

Compound Number : GSK1325760

Effective Date : 14-JAN-2020

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205019
- This RAP is intended to describe the analyses for primary and secondary endpoints required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Author | Date |
|---------------------------------------------|-------------|
| Manager (CPMS) | 24-OCT-2019 |
| Associate Statistician (FPD, Biostatistics) | 18-OCT-2019 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals (Method: E-mail):**

| Approver | Date |
|--------------------------------------------------------------|-------------|
| Project Statistician (FPD, Biostatistics) | 22-OCT-2019 |
| Study Accountable Person (Operations and Science Lead, GCSD) | 25-OCT-2019 |
| Medical Monitor (Clinical Sciences) | 22-OCT-2019 |
| DQL (Global Clinical & Data Operations) | 29-OCT-2019 |
| Senior Director (CPMS) | 23-OCT-2019 |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF e-signature):

| Approver | Date |
|-----------------------------------------------|-------------|
| Statistics Line Manager (FPD, Biostatistics) | 13-JAN-2020 |
| Programming Line Manager (FPD, Biostatistics) | 14-JAN-2020 |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | <mark>5</mark> |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s). Study Design Statistical Hypotheses / Statistical Analyses | 5<br>6 |
| 3. | PLANI<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | <mark>7</mark> |
| 4. | ANAL`<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING 'ENTIONS | 9 |
| 6. | STUD'<br>6.1.<br>6.2. | Y POPULATION ANALYSES Other Considerations for Data Analyses and Data Handling Conventions Overview of Planned Study Population Analyses | 10 |
| 7. | SAFE <sup>-</sup><br>7.1.<br>7.2.<br>7.3. | TY ANALYSESAdverse Events Analyses | 11<br>11 |
| 8. | PHAR<br>8.1. | MACOKINETIC ANALYSES Primary Pharmacokinetic Analyses 8.1.1. Endpoint / Variables 8.1.1.1. Drug Concentration Measures 8.1.2. Derived Pharmacokinetic Parameters 8.1.2. Summary Measure 8.1.3. Strategy for Intercurrent (Post Randomization) Events 8.1.4. Population of Interest 8.1.5. Statistical Analyses / Methods 8.1.5.1. Statistical Methodology Specification | 12<br>12<br>12<br>13<br>13<br>14 |
| 9. | REFEI | RENCES | 16 |
| 10. | APPEI<br>10.1.<br>10.2. | NDICES | 17<br>18 |

| | 10.2.2. | Screening and Follow-up Schedule of Events | 18 |
|---|---|---|---|
| | 10.2.3. | Treatment Periods 1, 2 and 3 (minimum of 7 days | |
| | | washout between doses) | 19 |
| 10.3. | | x 3: Assessment Windows | <mark>21</mark> |
| 10.4. | | x 4: Study Phases and Treatment Emergent Adverse | |
| | Events | | |
| | 10.4.1. | Study Phases | <mark>22</mark> |
| | | 10.4.1.1. Study Phases for Concomitant Medication | <mark>22</mark> |
| | 10.4.2. | Treatment Emergent Flag for Adverse Events | <mark>22</mark> |
| 10.5. | Appendix | x 5: Data Display Standards & Handling Conventions | <mark>23</mark> |
| | 10.5.1. | Reporting Process | <mark>23</mark> |
| | 10.5.2. | Reporting Standards | <mark>23</mark> |
| | 10.5.3. | Reporting Standards for Pharmacokinetic | <mark>24</mark> |
| 10.6. | Appendix | x 6: Derived and Transformed Data | 25 |
| | 10.6.1. | General | 25 |
| | 10.6.2. | Study Population | 25 |
| | 10.6.3. | Safety | 26 |
| | 10.6.4. | Pharmacokinetic | 26 |
| 10.7. | Appendix | x 7: Reporting Standards for Missing Data | <mark>27</mark> |
| | 10.7.1. | Premature Withdrawals | |
| | 10.7.2. | Handling of Missing Data | 27 |
| | | 10.7.2.1. Handling of Missing and Partial Dates | 27 |
| 10.8. | Appendix | x 8: Values of Potential Clinical Importance | 29 |
| | 10.8.1. | Laboratory Values | 29 |
| | 10.8.2. | | |
| | 10.8.3. | Vital Signs | 30 |
| 10.9. | Appendix | x 9: Abbreviations & Trade Marks | |
| | 10.9.1. | Abbreviations | 31 |
| | 10.9.2. | Trademarks | 32 |
| 10.10 | Appendix | x 10: List of Data Displays | |
| | | Data Display Numbering | |
| | 10.10.2 | Mock Example Shell Referencing | |
| | 10.10.3 | Deliverables | |
| | 10.10.4 | Study Population Tables | |
| | 10.10.5 | Safety Tables | |
| | 10.10.6 | Safety Figures | |
| | 10.10.7 | Pharmacokinetic Tables | |
| | | Pharmacokinetic Figures | |
| | | ICH Listings | |
| | | Non-ICH Listings | |
| 10 11 | | x 11: Example Mock Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 2017N346964\_00.

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 21/Jun/2019).

Note: Although all PK parameters are included in the primary endpoints, only AUC and Cmax will be analysed by statistics in line with success definition in the protocol and the rest PK parameters will be reported and treated as of secondary importance.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the relative bioavailability of Ambrisentan (AMB 1 mg x 5 tablets) administered as tablets dispersed in water or administered orally, with marketed Ambrisentan (AMB 5 mg x 1 tablet) in healthy adult participants under fasted conditions | <ul> <li>Plasma pharmacokinetic parameters of AMB as data permits: Maximum observed plasma concentration (C<sub>max)</sub>, Time to Cmax (t<sub>max)</sub>, Area under concentration-time curve from time zero (predose) extrapolated to infinite time(AUC (0-∞)), area under the concentration-time curve from time zero (predose) to last time of quantifiable concentration AUC (0-t) and Terminal phase half-life (t<sub>½.)</sub>, time of last quantifiable concentration (t<sub>last</sub>)</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To monitor the safety and tolerability of Ambrisentan (AMB 1 mg x 5 tablets) administered as tablets dispersed in water or administered orally, compared with marketed Ambrisentan (AMB 5 mg x 1 tablet) administered orally, in healthy adult | Adverse events (AE), vital signs, electrocardiogram (ECG), and clinical laboratory values. |
| Exploratory Objectives | Exploratory Endpoints |
| <ul> <li>To investigate palatability of AMB (1<br/>mg x 5 tablets) dispersed in water, in<br/>healthy adult participants.</li> </ul> | Palatability questionnaire scores |

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

This is an investigative study to study the pharmacokinetic parameters of a new formulation of AMB. Due to its descriptive nature, there will be no formal statistical hypothesis tested.

An estimation approach will be used to i) estimate the bioavailability of the test formulation relative to the reference formulation, and ii) for AUC (0-inf), AUC(0-t) and Cmax, point estimates and corresponding 90% confidence intervals will be constructed for the ratio of the geometric mean of the test formulation to the geometric mean of the reference formulation.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No Interim Analysis is planned for this study

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. Randomization codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | <b>Analyses Evaluated</b> |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Screen failures</li> </ul> |
| Randomized • All participants who were randomly assigned to treatment in the study. • This population will be based on the treatment the participant was randomized to. | | Study Population |
| Safety | All randomized participants who take at least 1 dose of study intervention. Participants will be analysed according to the intervention they actually received. | Safety Population |
| Pharmacokinetic<br>Concentration (PK) | The PK Concentration Population will include all participants for whom at least one PK sample was obtained and analysed. | • PK |
| Pharmacokinetic<br>Parameter<br>(PK_PAR) | For each PK parameter, the PK Parameter Population will include all participants who provide PK parameter data. | PK_PAR |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan final version, 27-SEP-2019.

- Data will be reviewed prior to Database Release (DBR) to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the electronic case report form eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

Treatment comparisons will be displayed as follows using the descriptors as specified:

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| F1 | GSK1325760 5 mg dispersed in water | Dispersed GSK1325760 | 1 |
| F2 | GSK1325760 5 mg administered orally | Oral GSK1325760 | 2 |
| R | Marketed AMB | Marketed AMB | 3 |

- 1. Dispersed GSK1325760 vs Marketed AMB (F1 vs R)
- 2. Oral GSK1325760 vs Marketed AMB (F2 vs R)

Note: Relevant footnotes to be added in all the displays as:

Dispersed GSK1325760: 5 mg (5 x 1 mg tablets) AMB tablet dispersed in water

Oral GSK1325760: 5 mg (5 x 1 mg tablets) AMB tablet administered orally

Marketed AMB: 5 mg (1 x 5 mg tablet) AMB tablet administered orally

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | • | |
| Vital Signs | X[1] | | X[1] | Day 1 (mean of the pre-dose)[2] |
| ECG | X[1] | | X[1] | Day 1 (worst case pre-dose)[2] |
| Haematology+ Clinical<br>Chemistry +<br>Urinalysis <sup>[3]</sup> | Х | Х | | Day-1 |

#### NOTES:

- [1] Taken in triplicate
- [2] Worst case of the triplicate pre-dose assessments for ECG will be the maximum value of the three measurements for each of the ECG parameter and mean of the pre-dose for Vital signs
- [3] Urinalysis baseline value required only when microscopic examination done

#### 6. STUDY POPULATION ANALYSES

# 6.1. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Reporting Standards for Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |

## 6.2. Overview of Planned Study Population Analyses

The study population analyses will be based on the randomized population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 8. PHARMACOKINETIC ANALYSES

## 8.1. Primary Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic Concentration (PK)" population, unless otherwise specified.

Table below provides an overview of the planned analysis, with the full details being presented in Appendix 10: List of Data Displays:

| Display Type | Untransformed | | | | | | | Ln-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | Summary | | Individual | | Stats Analysis | | lysis | Summary | | Individual | | |
| | T | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| PK Concentrations | | | | Y | Y[1] | Y[1] | Y | | | | | | | |
| Plasma PK<br>Parameters | Υ | | | Υ | Y[1] | Υ | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- . Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. [1] Linear and Semi-Logarithmic plots will be created on the same display.
- 2. [2] Separate mean and median plots will be generated.

## 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Standards for Pharmacokinetic)

Concentrations of ambrisentan in plasma will be listed and summarised by treatment and actual time.

Standard summary statistics will be calculated (i.e. arithmetic mean, standard deviation, median, minimum and maximum).

Refer to the PK Guidance document, titled Non-Compartmental Analysis of Pharmacokinetic Data (GUI\_51487) for more information regarding the treatment of concentrations below the assay's lower limit of quantification (NQ).

Individual plasma concentration-time profiles and median/mean profiles by treatment will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the loge-transformed scale (i.e., log-linear plot). In addition, a plot showing all individual subjects for each treatment will be produced (both linear and log-linear).

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin [version 8.1 or above]. All

calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters will be determined from the plasma concentration-time data, as data permits, for each subject and treatment unless otherwise specified. If parameters cannot be determined, a flag will be present in the data.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last |
| | quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for |
| | each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-inf) | Area under the concentration-time curve extrapolated to infinity will be calculated as: |
| | AUC(0-inf) = AUC(0-t) + Ct / lambda_z |
| | where Ct is the last observed quantifiable concentration. |
| Cmax | Maximum observed concentration determined directly from the concentration-time data. |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t1/2* | Apparent terminal half-life will be calculated as: |
| | t1/2 = In2 / lambda_z |
| %AUCext | The percentage of AUC(0-∞) obtained by extrapolation (%AUCex) will be calculated |
| | as: |
| | [AUC(0-∞) – AUC(0-t)] / AUC(0-∞) x 100 |
| Ct | The last observed quantifiable concentration |
| Tlast | Time of last quantifiable concentration |
| * associate | d parameters lambda_z, lambda_z_lower, lambda_x_upper, No_points_lambda_z to be listed. |
| NOTES: | |
| Additional paran | Additional parameters may be included as required. |
| Lambda_z is the | terminal phase rate constant. |

Derived pharmacokinetic parameters will be listed by subject and treatment. Listings will also include the individual subject ratios for AUC(0-inf), AUC (0-t) and Cmax, and the first point, last point and number of points used in the determination of  $\lambda z$ .

## 8.1.2. Summary Measure

- For each of the parameters AUC (0-inf), AUC (0-t), t1/2 and Cmax, the following summary statistics will be calculated and tabulated by treatment:
  - **Untransformed Data**: N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum
  - Loge-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of loge-transformed data and %CVb

For tmax, the summary statistics specified for untransformed data above will be generated.

As per the intercurrent events observed as defined in Section 8.1.3, relevant datapoints will be excluded from the pharmacokinetic parameters summary tables.

• Relative bioavailability of the new formulation of AMB and referenced or marketed AMB will be analysed by using AUC(0-t), AUC (0-∞), Cmax parameters

#### 8.1.3. Strategy for Intercurrent (Post Randomization) Events

Participants who experienced the following intercurrent events will have data from the relevant treatment period excluded from analysis:

- Did not receive full dosing
- Had a vomit within the first 2.5 hours after dose completion
- Did not provide an adequate PK concentration profile to allow reliable estimation of PK parameters

#### 8.1.4. Population of Interest

The primary statistical analyses will be based on the Pharmacokinetic parameter population (PK\_PAR), unless otherwise specified.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

### **Endpoint / Variables**

Log<sub>e</sub>-transformed AUC<sub>(0-t)</sub>, AUC <sub>(0-∞)</sub>, C<sub>max</sub> PK parameters of test formulation of GSK1325760 (F1, F2) and marketed AMB (R)

#### **Model Specification**

- Will be statistically analyzed separately using a mixed model (MM) for all treatment periods
- Terms fitted in the mixed effect ANOVA model will include:
  - o Fixed Effect: Treatment (F1, F2, R), Treatment Period
  - Random Effect: Subject
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used
- Point estimates for the adjusted means on the log<sub>e</sub> scale, the mean difference between treatments and associated 90% confidence interval for the contrast (test-reference) will be constructed using the residual variance for the following differences of interest:
  - AMB (1 mg x 5 tablets) administered as tablets dispersed in water(F1) and administered orally(F2) versus marketed AMB (R)(5 mg x 1 tablet) administered orally
- As per the observed intercurrent events, the strategy in sec 8.1.3 will be followed to exclude data points following the definition of intercurrent events

#### **Model Checking & Diagnostics**

For the Mixed Model analysis, Model assumptions will be applied, but appropriate adjustments may be made based on the data.

- Distributional assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model respectively) to
  gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared, or square root of data, will be explored

#### **Model Results Presentation**

- The point estimate and confidence interval obtained from MM analysis will be exponentially back-transformed to obtain Adjusted (least square) geometric means for each treatment
- Point estimates (Relative Bioavailability of GSK1325760) and associated 90% confidence interval for the ratio F1/R and F2/R along with within-subject variability (%CV<sub>w</sub>) will be reported Where
  - %CV<sub>w</sub>=100\*(SQRT (EXP( $\sigma_w^2$ )-1)) and  $\sigma_w^2$  is the mean squares error (MSE) from the statistical Mixed model
- Geometric Mean along with 90% CI treatment Ratios of GSK1325760 Plasma Derived Pharmacokinetic Parameters will also be plotted as in Section 10.10.8

## 9. REFERENCES

GlaxoSmithKline Document Number 2017N346964\_00: An open-label, randomized three period cross-over relative bioavailability study to compare the pharmacokinetic parameters of a lower dose formulation of ambrisentan (GSK1325760) with marketed ambrisentan in healthy adult participants.

## 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

A Per Protocol Population is not being defined for this study. Please Refer to Section 4.1 for handling and Reporting of Protocol Deviations.

## 10.2. Appendix 2: Schedule of Activities

## 10.2.1. Protocol Defined Schedule of Events

## 10.2.2. Screening and Follow-up Schedule of Events

| Procedure | Screening <sup>1</sup><br>(up to 28 days<br>before first dose) | Follow up/Early<br>Withdrawal<br>(7-14 days post<br>last dose) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Inclusion and exclusion criteria | X | | |
| Demography | X | | |
| Medical history (includes substance usage) | X | | Substances: Drugs, Alcohol, tobacco |
| Full physical exam, including height and weight | X | | |
| Brief physical exam | | Χ | |
| HIV, Hep B and Hep C screen | Х | | |
| Clinical chemistry,<br>haematology and urinalysis | X | Х | Only screening tests need to be fasted |
| FSH | Х | | Required only in women to confirm postmenopausal status |
| Alcohol breath test | Х | | |
| Urine or serum drugs test | X | | |
| Vital signs (blood pressure, heart rate and temperature) | X | Х | Triplicate blood pressure and heart rate required at screening. |
| 12-lead ECG | Х | Х | Triplicate ECG required at screening. |
| Concomitant Medication review | Х | Х | Con meds before dosing can be recorded in medical history |
| AE/SAE review | X | X | Refer to protocol Section 8.3.1 |

<sup>1.</sup> Screening assessments may be conducted at multiple visits, if required.

## 10.2.3. Treatment Periods 1, 2 and 3 (minimum of 7 days washout between doses)

| | | | | | | Day | y 1 (ho | urs) | Day 2 | | Day 3 Day 4 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day -1 | Pre-<br>dose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 4 | 8 | 12 | 18 | 24 | 36 | 48 | 72 | Notes |
| Clinic Visits | | | | | | | | | | | | | | | | | |
| Out-patient Visit | | | | | | | | | | | | | | | | Х | |
| Admission to clinic | Х | | | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | | | | | x | | If more convenient for participants, they can remain in the unit until 72 h, at the discretion of the investigator |
| Study Intervention | | | | | | | | | | | | | | | | | |
| Randomisation | | Х | | | | | | | | | | | | | | | Can be done on Day –1 or<br>Pre-dose Day 1. Only in<br>Treatment Period 1 |
| Study Intervention | | | Х | | | | | | | | | | | | | | Fasted from midnight until 4<br>h afterwards, except for<br>water, allowed ad libitum,<br>except for 1 h before and<br>after dosing |
| Safety Assessments | | | | | | | | | | | | | | | | | |
| Vital signs (blood pressure, heart rate and temperature) | | Χ | | Χ | Χ | | Χ | | Х | Χ | Х | | Х | | Χ | Χ | Triplicate pre-dose. Single measurements at other |
| 12-lead ECG | | Х | | | Х | | Х | | х | | х | | Х | | | Х | timepoints, unless out of<br>range, then triplicates<br>should be performed |
| Clinical chemistry, haematology and urinalysis | Х | | | | | | | | | | | | | | Х | | Fasting not required |
| Brief physical examination | Х | | | | | | | | | | | | | | | | |

| | | | Day 1 (hours) | | | | | | | | | | | | | Day 4 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day -1 | Pre-<br>dose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 4 | 8 | 12 | 18 | 24 | 36 | 48 | 72 | Notes |
| Alcohol breath test | Х | | | | | | | | | | | | | | | | |
| Urine or serum drugs test | Х | | | | | | | | | | | | | | | | |
| Concomitant Medication | Х | х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Con meds before dosing can be recorded in medical history |
| SAE/AE review | <b>◄===</b> | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | | ===== | | ===== | | ===== | == <b>&gt;</b> | Refer to Protocol Section 8.3.1 |
| Other Assessments | | | | | | | | | | | | | | | | | |
| PK blood samples | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Platability Questionnaire | | | X | | | | | | | | | | | | | | Questionnaire only to be completed in the Treatment Period dosing AMB tablets dispersed in water. To be completed within 10 min of dosing |

- When scheduled at the same time-points, 12-lead ECGs and vital signs should be completed before any blood draws.
- The timing of assessments should allow PK samples to be taken as close as possible to the nominal time-point.
- The timing and number of planned safety assessments and pharmacokinetic samples may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files but will not constitute a protocol amendment. The Competent Authority (CA) and ethics committee (EC) will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the informed consent form (ICF). The changes will be approved by the CA and the EC before implementation.

## 10.3. Appendix 3: Assessment Windows

Required assessment windows are specified in the Study Reference Manual for this study.

# 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 10.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment.

#### 10.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior, and up to the last scheduled visit |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 10.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date. (plus, washout or protocol-specified time limit (e.g. half-life of drug, certain number of days, etc.).</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date+ 1 day</li> <li>If AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period: Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date+ 1 day </li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Reporting Process

| Software | Software |
|---|---|
| The SAS Version | 9.4 or above and WinNonlin Version 8.1 or above will be used. |
| Reporting Area | |
| HARP Server : uk1salx00175 | |
| HARP Compound | : dmwork/gsk1325760/mid205019 |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets will be created according to latest IDSL | |
| Generation of RTF Files | |
| RTF files will be g | enerated for final SAC |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx)
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N. n. frequency, % |

| Gr | Graphical Displays |
|----|----------------------------------------------------|
| • | Refer to IDSL Statistical Principals 7.01 to 7.13. |

## 10.5.3. Reporting Standards for Pharmacokinetic

| Reporting of Pharm | nacokinetic Concentration Data |
|---|---|
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary Statistics | Refer to IDSL Statistical Principle 6.06.1. |
| | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Reporting of Pharm | nacokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between and or within geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> <li>[2] CV<sub>w</sub> (%) = √ (exp(MSE) - 1) * 100 (MSE = mean square error from mixed effect model of loge-transformed data).</li> </ul> |
| Parameters Not<br>Being Log<br>Transformed | $T_{\text{max}}$ , $T_{\text{last}}$ , first point, last point, and number of points used in the determination of $\lambda z$ , %AUCex |
| Summary Tables | All provided PK parameters will be summarised except Lamz, lamzUL, LamzLL, LamzNP and AUC % extrapolated area , Rsq-adjusted (if calculated). |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### **Palatability Questionnaire**

Time difference between dose and questionnaire will be derived as:
 Date/time of assessment - Date/time of dose

If this difference <= 10 min, then this subject will be flagged as Y else N A separate flag variable for particularly this treatment will record value as Y or N

#### 10.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
- Since Year of Birth is recorded in eCRF, date and month will be imputed as '30th June' of that Year.
  - Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

 Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.

#### 10.6.3. Safety

#### **Laboratory Parameters**

If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

- Example 1: 2 Decimal Places = '< x' becomes x 0.01</li>
- Example 2: 1 Decimal Places = '> x' becomes x + 0.1
- Example 3: 0 Decimal Places = '< x' becomes x − 1

#### **Adverse Events**

#### **AE'S OF Special Interest**

Not Applicable

#### ECG Parameters

• Machine read values of PR, QRS, QT, QTc, QTcB, QTcF will be captured

#### 10.6.4. Pharmacokinetic

## **PK Endpoints**

• Not required in this section, please refer Section 8.1

## 10.7. Appendix 7: Reporting Standards for Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as A participant is considered to have completed the study if he/she has completed all phases of the study including the follow-up visit. |
| | Withdrawn participants will not be replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be summarised as withdrawal visits. |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/ | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |

| Element | Reporting Detail |
|---|---|
| Medical | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be</li> </ul> |
| History | used for the month |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent<br/>on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.8. Appendix 8: Values of Potential Clinical Importance

## 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Datio of | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | ı | $\Delta$ from BL | > 0.075 | |
| | ~/I | Male | | 180 |
| Haemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | >25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | >44.2 |
| Glucose (fasting at screening) | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| BUN | mmol/L | | | 2x ULN (mmol/L) |
| Liver Function | | | | |
| Test Analyte | Units | Category | Clinical Concern Range | |
| ALT/SGPT | U/L | High | >=2xULN | |
| AST/SGOT | U/L | High | >=2xULN | |
| AlkPhos | U/L | High | >=2xULN | |
| T Bilirubin | µmol/L | High | >=1.5xULN | |

## 10.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | 500 |
| Absolute PR Interval | msec | 110 | 220 |
| Absolute QRS Interval | msec | 75 | 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

## 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | 85 | 160 |
| Diastolic Blood Pressure | mmHg | 40 | 110 |
| Heart Rate | bpm | 45 | 100 |

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Change from Baseline) | | Increase | |
| | | Lower | Upper |
| Systolic Blood Pressure | mmHg | | >30 |
| Diastolic Blood Pressure | mmHg | | >20 |

## 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| AUC(0-inf) | Area under the concentration-time curve from time zero (predose) extrapolated |
| , | to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (predose) to time of last |
| | quantifiable concentration within a participant across all treatments |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| NQ | Non-quantifiable |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |

| Abbreviation | Description |
|---|---|
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SD | Standard deviation |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| tlag | Lab time before observation of drug concentrations in sampled matrix |
| tlast | Time of last quantifiable concentration |
| tmax | Time of occurrence of Cmax |
| WNL | Windows Non Linear |

## 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ADVAIR |
| HARP |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin 8.1 or above |

## 10.10 Appendix 10: List of Data Displays

#### 10.10.1 Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.11 | N/A |
| Safety | 3.1 to 3.23 | 3.1 to 3.2 |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 to 4.6 |
| Section | Listi | ngs |
| ICH Listings | 1 to 26 | |
| Other Listings | 27 to 32 | |

All displays (Tables, Figures & Listings) will use the term 'Subjects'.

## 10.10.2 Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|---------|---------|
| Study Population | NA | POP_T1 | NA |
| Safety | NA | SAFE_T1 | SAFE_L1 |
| Pharmacokinetic | PK_F1 | NA | NA |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3 Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| DR | Dry Run |
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.10.4 Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of subject Disposition for the subject Conclusion Record | ICH E3, FDAAA, EudraCT | DR, SAC |
| 1.2. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | DR, SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | DR , SAC |
| 1.4. | Screened | NS1 | Summary of Number of subjects by Country and Site ID | EudraCT/Clinical Operations | DR, SAC |
| Populati | on Analysed | | | | • |
| 1.5. | Screened | SP1 | Summary of Study Populations | IDSL | DR , SAC |
| Demogra | aphic and Basel | ine Characteristic | CS CS | | |
| 1.6. | Safety | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | DR, SAC |
| 1.7. | Randomized | DM11 | Summary of Age Ranges | EudraCT | DR, SAC |
| 1.8. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | DR , SAC |
| Prior and | d Concomitant I | Medications | | | • |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.9. | Safety | MH1 | Summary of Current/Past Medical Conditions | ICH E3 | DR, SAC |
| Palatability | Palatability Questionnaire | | | | |
| 1.10 | Safety | POP_T1 | Responder's Summary of Palatability Questionnaire | Non-standard | DR, SAC |
| 1.11 | Safety | SAFE_T1 | Responder's compliance to 10 mins for Palatability Questionnaire | Non-standard | DR, SAC |

# 10.10.5 Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events (AEs) | | | | |
| 3.1. | Safety | AE1CP | Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term | ICH E3 | DR , SAC |
| 3.2. | Safety | AE1CP | Summary of Treatment Emergent Drug-Related Adverse Events by System Organ Class and Preferred Term/by Overall Frequency | ICH E3 | DR , SAC |
| 3.3. | Safety | AE15 | Summary of Common (>=2%) Non-serious Treatment Emergent<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | FDAAA, EudraCT | DR , SAC |
| Serious | Serious and Other Significant Adverse Events | | | | |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.4. | Safety | AE16 | Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Number of subjects and Occurrences) | FDAAA, EudraCT | DR , SAC |
| 3.5. | Safety | CP_AE1x | Summary of Treatment Emergent Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency | IDSL | DR , SAC |
| Labora | tory: Chemistry | y | | | |
| 3.6. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | DR , SAC |
| 3.7. | Safety | LB1 | Summary of Chemistry Values | | DR, SAC |
| 3.8. | Safety | LB17 | Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | DR , SAC |
| Labora | tory: Hematolo | ду | | | • |
| 3.9. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | DR , SAC |
| 3.10. | Safety | LB1 | Summary of Hematology Values | | DR, SAC |
| 3.11. | Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | DR , SAC |
| Labora | tory: Urinalysis | 3 | | | |
| 3.12. | Safety | UR1 | Summary of Worst-Case Urinalysis Results Post-Baseline Relative to Baseline | ICH E3 | DR , SAC |
| Safety: | Tables | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL / Example Shell Title Programming Notes | | Programming Notes | Deliverable<br>[Priority] | |
| 3.13. | Safety | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 Only where microscopic examination is done | DR , SAC | |
| Labora | tory: Hepatobil | iary (Liver) | | | | |
| 3.14. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | DR, SAC | |
| 3.15. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | DR, SAC | |
| ECG | | 1 | | | 1 | |
| 3.16. | Safety | EG1 | Summary of ECG Findings | IDSL | DR , SAC | |
| 3.17. | Safety | EG2 | Summary of ECG Values | IDSL | DR, SAC | |
| 3.18. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL | DR, SAC | |
| 3.19. | Safety | CP_EG9 | Summary of Change from Baseline in ECG Values by Visit | IDSL | DR, SAC | |
| 3.20. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | IDSL | DR, SAC | |
| Vital Si | gns | 1 | | | 1 | |
| 3.21. | Safety | VS1 | Summary of Vital Signs | IDSL All vital signs including heart rate and temperature to be summarised. | DR, SAC | |
| 3.22. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 All vital signs including heart rate and temperature to be summarised. | DR , SAC | |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.23. | Safety | VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | IDSL | DR , SAC |

# 10.10.6 Safety Figures

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title | | | Programming Notes | Deliverable<br>[Priority] |
| Laborat | Laboratory | | | | |
| 3.1. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | IDSL | DR , SAC |
| 3.2. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | IDSL | DR , SAC |

## 10.10.7 Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title Programming Notes | | Deliverable<br>[Priority] |
| Plasma | GSK1325760 | | | | |
| 4.1. | PK | Pkct1 | Summary of Plasma GSK1325760 Concentration-Time data by treatment | | DR , SAC |
| 4.2. | PK_PAR | Pkpt1 | Summary of Untransformed Plasma GSK1325760 Derived Pharmacokinetic Parameters by treatment | Parameters with units | DR , SAC |
| 4.3. | PK_PAR | Pkpt3 | Summary of Loge-transformed Plasma GSK1325760 Derived Pharmacokinetic Parameters by treatment | Parameters with units | DR , SAC |
| PK Stat | PK Statistical Analysis | | | | |
| 4.4. | PK_PAR | PK_T1 | Summary of Statistical Analysis of Loge-transformed Plasma GSK1325760 Derived PK Parameters | Footnotes as in example mock shell by treatment | DR , SAC |

# 10.10.8 Pharmacokinetic Figures

| Pharma | acokinetic: Figu | ıres | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Plasma | GSK1325760 | | | | |
| 4.1. | PK | Pkcf6 | Individual Subject Plasma GSK1325760 Concentration-Time Plots (Linear and Semi-log) by Treatment | Spaghetti plots, all subjects by treatment. | DR, SAC |
| 4.2. | PK | Pkcf1x | Individual Subject GSK1325760 Plasma Concentration-Time Plot (Linear and Semi-log) by Subject | Paginate by Subject. Different point symbol (and colour) to be used for each treatment and to be mentioned in footnote of the figure. | DR, SAC |
| 4.3. | PK | Pkcf4 | Arithmetic Mean(+SD) GSK1325760 Concentration-Time Plots (Linear and Semi-log) by Treatment | Different line type (and colour) to be used for each treatment and to be mentioned in footnote of the figure All treatments on one page. | DR, SAC |
| 4.4. | PK | Pkcf5 | Median(range) Plasma GSK1325760 Concentration - time Plot (Linear and Semi-log) by Treatment | Different line type (and colour) to be used for each treatment and to be mentioned in footnote of the figure All treatments on one page. | DR, SAC |
| 4.5. | PK_PAR | Pkpf3 | Comparative Plot of Individual Subject GSK1325760 Plasma Concentration-Time Derived Parameters vs. Treatment (Linear and semi-logarithmic) | Needed for only AUC(0-inf), AUC(0-t) and Cmax, each parameter on different page. For each parameter all treatments on one page. | DR, SAC |
| 4.6. | PK_PAR | PK_F1 | Geometric Mean (90% CI) Treatment Ratios of GSK1325760 Plasma Derived Pharmacokinetic Parameters | Comparison F1-R, F2-R. Needed for only AUC(0-inf), AUC(0-t) and Cmax. [Non-Standard] | DR, SAC |

# 10.10.9 ICH Listings

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | • |
| 1. | Safety | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | DR , SAC |
| 2. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | DR , SAC |
| Protoc | ol Deviations | , | | | • |
| 3. | Safety | DV2A | Listing of Important Protocol Deviations | ICH E3 | DR , SAC |
| 4. | Safety | IE4 | Listing of subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | DR, SAC |
| Demog | raphic and Bas | eline Characteris | tics | | • |
| 5. | Safety | DM4 | Listing of Demographic Characteristics | ICH E3 | DR, SAC |
| 6. | Safety | DM10 | Listing of Race | ICH E3 | DR, SAC |
| Prior a | nd Concomitan | t Medications | | | • |
| 7. | Safety | CM5 | Listing of Concomitant Medications | IDSL | DR , SAC |
| Expos | ure and Treatme | ent Compliance | | | 1 |
| 8. | Safety | EX4 | Listing of Exposure Data | ICH E3 | DR, SAC |
| Advers | se Events | | | | |
| 9. | Safety | AE9CP | Listing of All Adverse Events | ICH E3 | DR, SAC |
| 10. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | DR, SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 11. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | DR , SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 12. | Safety | CP_AE9a | Listing of Fatal Serious Adverse Events | ICH E3 | DR , SAC |
| 13. | Safety | CP_AE9a | Listing of Non-Fatal Serious Adverse Events | ICH E3 | DR , SAC |
| 14. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | DR, SAC |
| 15. | Safety | CP_AE9 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | DR , SAC |
| All Lab | oratory | | | • | |
| 16. | Safety | CP_LB6 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance/Outside Normal Range | ICH E3 | DR , SAC |
| 17. | Safety | CP_LB6 | Listing of Laboratory Values of Potential Clinical Importance | | DR, SAC |
| 18. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | DR, SAC |
| 19. | Safety | UR2B | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 Abnormal dipstick findings and microscopic results | DR , SAC |
| ECG | | | | | |
| 20. | Safety | CP_EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | DR, SAC |
| 21. | Safety | CP_EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL | DR, SAC |
| 22. | Safety | CP_EG6 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL | DR, SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | Safety | CP_EG6 | Listing of Abnormal ECG Findings | IDSL | DR, SAC |
| Vital Sig | gns | | | | |
| 24. | Safety | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | DR, SAC |
| 25. | Safety | CP_VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL | DR, SAC |
| 26. | Safety | CP_VS5 | Listing of CFB in Vital Signs of Potential Clinical Importance | IDSL | DR, SAC |

# 10.10.10 Non-ICH Listings

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Fitle Programming Notes | | Deliverable<br>[Priority] |
| PK | | | | | |
| 27. | PK | pkcl1x | Listing of Plasma GSK1325760 Concentration-time Data by treatment | List all the concentration data including unscheduled | DR, SAC |
| 28. | PK_PAR | pkpl1p | Listing of Derived Plasma GSK1325760 Pharmacokinetic Parameters by Treatment | | DR, SAC |
| 29. | PK_PAR | Pkpl2 | Listing of GSK1325760 Pharmacokinetic Parameter Ratios by treatment | | DR, SAC |
| 30. | PK_PAR | NA | RAW SAS Output from Statistical Analysis of GSK1325760 Plasma Pharmacokinetic Parameters | | DR, SAC |
| Study F | opulation | | | | |
| 31. | Safety | SAFE_L1 | Listing of all subjects with the time of answering palatability questionnaire | Footnotes | DR, SAC |

## 10.11 Appendix 11: Example Mock Shells for Data Displays

Example: POP\_T1 Protocol: 205019 Population: Safety

Table 1.10 Responder's Summary of Palatability Questionnaire

 Question No.
 Dispersed GSK1325760 (N=20)

 Response
 n(%)



Note:
Question 1:
Question 2:
Question 3:

Dispersed GSK1325760 : 5 mg (5 x 1 mg tablets) AMB tablet dispersed in water

Example: SAFE\_T1 Protocol: 205019 Population: Safety

Table 1.11
Responder's compliance to 10 mins for Palatability Questionnaire

| Treatment Period | Dispersed GSK1325760<br>(N=8)<br>n(%) |
|------------------|---------------------------------------|
| Period 1 | 4(50%) |
| Period 2 | 8(100%) |
| Period 3 | 8(100%) |

Footnote:

Dispersed GSK1325760 : 5 mg (5 x 1 mg tablets) AMB tablet dispersed in water

2019N426492\_00 205019

Example : PK\_T1 Page 1 of n

Protocol: mid205019 Population: PK\_PAR

Table 4.4 Summary of Statistical Analysis of Loge-transformed Plasma GSK1325760 PK Parameters

| Parameter | Comparison<br>Test vs Reference | Adjusted Geome | tric Mean | Ratio<br>(Test/Ref) | 90% Confidence<br>Interval for the Ratio | %CVw |
|---|---|---|---|---|---|---|
| | rest vs releience | n Test n Ref | (16301XeI) | interval for the Natio | | |
| AUC(0-inf)(units) | Dispersed GSK1325760<br>vs Marketed AMB | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | XX.X |
| AUC(0-t)(units) | Oral GSK1325760<br>vs Marketed AMB | X XX.XX | X XX.XX | x.xxx | (x.xxxx, x.xxxx) | XX.X |

#### FOOTNOTE:

Dispersed GSK1325760: 5mg (5x 1 mg tablets) AMB tablet dispersed in water Oral GSK1325760: 5mg (5 x 1 mg tablets) AMB tablet administered orally Marketed AMB: 5 mg (1 x 5 mg tablet) AMB tablet administered orally

Example : SAFE\_L1 Page 1 of n

Protocol : mid205019 Population : Safety

Listing 32

Listing of all subjects with the time of answering palatability questionnaire

| Subj. | {Age(y)/<br>Sex/<br>Race} | Treatme nt Period/ | Date/Time of<br>Dosing | Date/Time of Questionnaire | |
|---|---|---|---|---|---|
| PPD | 36/<br>M/<br>Mixed Race | Period<br>1/<br>Dispersed<br>GSK132576 | xx-xx-xx<br>xx:xx:xx | xx-xx-xx<br>xx:xx:xx | Xxx |
| PPD | 33/<br>M/<br>Mixed Race | Period<br>2/<br>Dispersed<br>GSK132576 | xx.xx | xx-xx-xx<br>xx:xx:xx | Xxx |
| PPD | 24/<br>M/<br>Mixed Race | Period<br>3/<br>Dispersed<br>GSK132576 | xx.xx | xx-xx-xx<br>xx:xx:xx | xxx |

### FOOTNOTE:

Dispersed GSK1325760: 5mg (5x 1 mg tablets) AMB tablet dispersed in water

Example : PK\_F1
Protocol : mid205019
Population : PK\_PAR

Page 1 of n

Figure 4.6

Geometric Mean Treatment Ratio and 90% CI of Analyte Matrix PK Parameters



Note: A,B,C are test treatments(in this case F1 and F2) and R is the Reference treatment

#### FOOTNOTE:

Dispersed GSK1325760: 5mg (5x 1 mg tablets) AMB tablet dispersed in water Oral GSK1325760: 5mg (5 x 1 mg tablets) AMB tablet administered orally Marketed AMB: 5 mg (1 x 5 mg tablet) AMB tablet administered orally